CLINICAL TRIAL: NCT05556928
Title: Cancer and Aging Resilience Evaluation in Older Adults With Hematologic Malignancies: The CARE-Heme Registry
Acronym: CARE-Heme
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Noha Mohamed Sharafeldin, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300005372
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Amyloidosis; Plasma Cell Leukemia
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis; Leukemia, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — The purpose of the biospecimen collection is to support future investigations aimed at looking at biomarkers of frailty and aging and other new-onset comorbidities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this protocol is to create a registry of older (≥50 years old) patients with Hematologic Malignancies. Our main objectives include: To understand the prevalence of frailty and geriatric impairments among patients aged ≥50y and above diagnosed with a hematologic malignancy at UAB and to gather information that would lend support for future research in this vulnerable population.

DETAILED DESCRIPTION:
All participants will be invited to participate in a patient reported geriatric assessment questionnaire as well as an objective physical function testing. This includes the Short Physical Performance Battery (SPPB) that evaluates lower extremity performance and muscle strength assessment via hand grip dynamometer. Participants will also complete a 12 item modified version of PRO-CTCAE. This will be administered by trained research staff at the time of study enrollment. Repeat CARE instruments (Follow-up GA questionnaire and Physical Function test) will be administered after the baseline visit to measure changes in patient reported outcomes at 3 months, 6 months, and one year. A one-time blood or saliva sample will be requested and obtained at baseline or a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients are ≥50 years of age.
* Patients have a biopsy proven diagnosis of Hematologic Malignancy (Multiple Myeloma, AL Amyloidosis, Waldenstrom's Macrogloblunemia, Hodgkin Lymphoma, Non-Hodgkin Lymphoma, Myelodysplastic syndromes, Myeloproliferative Neoplasm, Acute/Chronic Myeloid Leukemia, Acute/Chronic Lymphoid Leukemia).
* Patients have appointments at UAB including if they are an inpatient or other clinic locations.

Exclusion Criteria:

* Individuals who are <50 years old.
* Patients who do not read and/or speak English will not be eligible for this study as many of the questionnaires are not validated in other languages. No exclusions will be made based on gender, ethnicity or race.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥50 years of age with a diagnosis of any Hematologic Malignancy having an appointment at any participating UAB entity.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Create the CARE-Heme Registry | 5 years
  To establish and maintain a well-annotated registry (to be called the 'CARE-Heme' Registry) of adults ≥50 years of age with a hematologic malignancy to improve our understanding of this vulnerable population.

SECONDARY OUTCOMES:
To administer a patient reported geriatric assessment and a brief objective physical assessment. | 5 years
  To measure the proportion of patients with overall and domain-specific geriatric impairments, the proportion of patients with Myopenia, and the proportion of patients with frailty.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirklin Clinic of UAB Hospital, Birmingham, Alabama, United States